CLINICAL TRIAL: NCT03698890
Title: Evaluation of Clinical Pathways for Patients With Hypertension on Follow-up in the Polyclinics
Brief Title: Primary Technology Enhanced Care in Hypertension
Acronym: PTEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Healthcare Group Polyclinics (Other Government)
Collaborators: Ministry of Health, Singapore (Other Government)
Responsible Party: Principal Investigator, Valerie Teo, Family Physician, Associate Consultant, Deputy Head, Ang Mo Kio Polyclinic, National Healthcare Group Polyclinics
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018/00785
Record Dates: First submitted 2018-10-01; First posted 2018-10-09 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Hypertension
Keywords: Hypertension; Telehealth; Primary care; Teamlet
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual care of 3 to 6-monthly clinic visit
- Intervention (Experimental): Network-based home blood pressure monitor (Fora P20b Blood Pressure Monitor) and telephone consult with care team
  Interventions: Device: Network-based home blood pressure monitor

INTERVENTIONS:
Device: Network-based home blood pressure monitor — A network-based home blood pressure monitor will be loaned to patients in the intervention group, who will be asked to monitor their blood pressure at least once every week using the network based home blood pressure monitor, which automatically uploads measured blood pressure readings to the portal for care managers (CM) to review blood pressure readings and provide updates to the patient on blood pressure control. If a patient's blood pressure is elevated, the CM can titrate medications over the phone and provide follow up tele-consultation and necessary treatment.
  Other Names: Fora P20b Blood Pressure Monitor
  Arms: Intervention

SUMMARY:
This study evaluates the impact of the use of a technology-enabled home blood pressure monitor amongst hypertensive patients in primary care. Half of the patients will receive the blood pressure monitor for home monitoring, while the other half will receive usual care at the polyclinic. The hypothesis is tele-monitoring along with nurse led tele-support and medical review (i.e. tele-treatment) can enhance primary care management of hypertension by improving patient outcomes and reducing health costs.

DETAILED DESCRIPTION:
A literature review on telemedicine in primary care indicated that tele-monitoring can enhance primary care management of hypertension (HT) by improving patient outcomes and reducing health costs. In addition, technology-enabled blood pressure (BP) self-monitoring interventions have even better BP control outcomes if (i) nurse led tele-support and (ii) medication review (i.e. tele-treatment) are added.

This study comprises 2 phases:

Phase 1: Intervention phase This will be an open label (unblinded), parallel, non-randomized, quasi-experimental study conducted within 1 study site. Patients who are under the care of 2 clinical teams, called teamlets (comprising 2 family physicians, a care coordinator and a care manager who is a nurse), will be recruited into the study.

Patients under the care of 1 teamlet will be allocated to the intervention group, while those under the care of the other teamlet will be allocated to the usual care group.

One key modality for this study will be the use of a network-based home blood pressure monitor to provide patient-led tele-monitoring for BP levels for patients in the intervention group. The monitor will be loaned to patients in the intervention group, who will be asked to monitor their blood pressure at least once every week using the network based home blood pressure monitor, which automatically uploads measured blood pressure readings to the MyHealthSentinel (MHS) portal for care managers (CM) in the teamlet to review blood pressure readings.

The network-based home blood pressure monitor will be used to enhance nurse-led tele-support in the following ways:

1. the CM will access the MHS portal to review the patient's blood pressure and provide updates to the patient on blood pressure control.
2. If a patient's blood pressure is elevated, using the established protocols, the CM can titrate medications over the phone and provide follow up tele-consultation and necessary treatment in 2 to 4 weeks to assess subsequent blood pressure levels and side effects. The titration of medication is part of usual care and is managed by the ordering physician. Patients will be contacted after dose titration to see whether his or her blood pressure has improved. The care manager will also use the same phone call to check whether patients followed the titrated medication dosage.

Patients in the usual care group will continue to be followed up and managed as per usual, there will be no additional clinical intervention provided to patients in this group.

At 6 months after recruitment into the study, the patients' clinical outcomes will be measured. Specific outcome variables are as follows:

(i) blood pressure after 6 months, (ii) Proportion of HT patients with controlled BP at each month and (iii) Time to BP control (only if medications review is done). The above variables will be extracted from Electronic Medical Records database, as well as the MHS portal to derive the above mentioned outcome variables along with additional variables to be extracted.

A questionnaire will be administered to both groups at the first study visit and at the visit after 6 months to survey patients on their sodium intake, quality of life, beliefs about medication, medication adherence, and satisfaction with the care provided.

Patients in both arms will receive reimbursement at the end of study participation.

Phase 2: Qualitative phase A sub-group of patients (control group and intervention group) and teamlet staff, will be invited to participate in one-to-one semi-structured in-depth interviews and/or focus group discussions (FGDs), to find out their experience with the managing blood pressure via telemonitoring or physical clinic visit. All interviews and FGDs will be audio-recorded and later transcribed. Transcripts will not contain any personal data. Field notes will be taken during the interviews and memos written after the completion of interview. Both deductive and inductive approaches will be adopted to analyze the collected data using elements of thematic analysis and constant comparison approaches.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patients with hypertension only, or hypertension and hyperlipidemia
* Patients who are cared for by teamlets
* Patients who are technology savvy and are able and willing to use telemedicine devices, or have a family member who is willing to assist in using telemedicine for blood pressure control
* Clinic teams who are directly involved in patient care

Exclusion Criteria:

* Patients who have cognitive impairment
* Pregnant patients
* Patients with hypertension and other chronic illnesses other than hyperlipidemia, such as diabetes.
* Patients with a history of ischemic heart disease, congestive heart failure, stroke, transient ischemic attack, atrial fibrillation and renal impairment.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure control | 6 months
  Change in systolic and diastolic blood pressure (in mmHg) after 6 months. Readings will be obtained monthly from the MHS portal.

SECONDARY OUTCOMES:
Time to blood pressure control | 6 months
  Trend of time taken for blood pressure to be controlled if medication review is done. Readings will be obtained monthly from the MHS portal. This will be measured in hours, days or months.
Proportion of participants with controlled blood pressure | 6 months
  Change in proportion of participants with controlled blood pressure, measured by systolic & diastolic blood pressure, at each month. This will be measured in percentage.
Healthcare utilization of participants | 6 & 12 months
  Trend of utilization of healthcare services by participants. These include number of hospitalizations, doctor consultations, nurse consultations, teleconsultations, treatment & procedures, screening, laboratory tests, pharmacy services. These information will be obtained from the electronic medical records.
Healthcare costs incurred by participants | 6 & 12 months
  Change in costs of healthcare services utilized by participants. These include administrative costs, costs of doctor consultations, nurse consultations, teleconsultations, treatment & procedures, medications, screening, laboratory tests, pharmacy services. These information will be obtained from institution's Finance system and the electronic medical records. All amounts will be in Singapore dollars.
Number of medications prescribed to participants | 6 months
  Change in number of medications prescribed to participants during the course of study participation. This information will be obtained from the electronic medical records.
Type of medications prescribed to participants | 6 months
  Change in type of medications prescribed to participants during the course of study participation, e.g. antihypertensive drug class. This information will be obtained from the electronic medical records.
Quality of life of participants | 6 months
  Change in quality of life of participants. This will be measured by the 5-level EuroQol 5-dimension questionnaire (EQ-5D-5L) which will be completed by participants at the baseline visit and 6-month phone call. The scale measures self-reported health outcomes. Each of the 5 domains will be coded from 1 to 5, and the final 5-digit health state will be converted into a single index value to facilitate calculation of quality-adjusted life years (QALY).
Medication adherence | 6 months
  Change in medication adherence of participants. This will be measured by self-report through a questionnaire with 4-point Likert scale, adapted from the Hill-Bone Compliance to High Blood Pressure Therapy Scale. Total score for each patient will be from 4 to 12, with higher scores reflecting poorer adherence to medication. This will be completed at the baseline visit and 6-month phone call.
Patient satisfaction | 6 months
  Patient satisfaction with telemonitoring or usual care will be measured by a self-reported questionnaire on a 6-point Likert scale which will be completed at the 6-month phone call. Total score for each patient will be from 6 to 30 with higher scores reflecting better satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Teo, Principal Investigator — National Healthcare Group Polyclinics
Locations (1):
- Ang Mo Kio Polyclinic, Singapore, Singapore

REFERENCES:
- [Background] Duan Y, Xie Z, Dong F, Wu Z, Lin Z, Sun N, Xu J. Effectiveness of home blood pressure telemonitoring: a systematic review and meta-analysis of randomised controlled studies. J Hum Hypertens. 2017 Jul;31(7):427-437. doi: 10.1038/jhh.2016.99. Epub 2017 Mar 23. PMID 28332506
- [Background] Purcell R, McInnes S, Halcomb EJ. Telemonitoring can assist in managing cardiovascular disease in primary care: a systematic review of systematic reviews. BMC Fam Pract. 2014 Mar 7;15:43. doi: 10.1186/1471-2296-15-43. PMID 24606887
- [Background] Chandak A, Joshi A. Self-management of hypertension using technology enabled interventions in primary care settings. Technol Health Care. 2015;23(2):119-28. doi: 10.3233/THC-140886. PMID 25515051
- [Background] Bosworth HB, Olsen MK, Grubber JM, Neary AM, Orr MM, Powers BJ, Adams MB, Svetkey LP, Reed SD, Li Y, Dolor RJ, Oddone EZ. Two self-management interventions to improve hypertension control: a randomized trial. Ann Intern Med. 2009 Nov 17;151(10):687-95. doi: 10.7326/0003-4819-151-10-200911170-00148. PMID 19920269
- [Derived] Teo SH, Chew EAL, Ng DWL, Tang WE, Koh GCH, Teo VHY. Implementation and use of technology-enabled blood pressure monitoring and teleconsultation in Singapore's primary care: a qualitative evaluation using the socio-technical systems approach. BMC Prim Care. 2023 Mar 16;24(1):71. doi: 10.1186/s12875-023-02014-8. PMID 36927496